CLINICAL TRIAL: NCT07388264
Title: Examining the Impact of Weizmannia (Bacillus) Coagulans JBI-YZ6.3 on Gut Health and Fecal Microbiome Changes
Brief Title: Impact of Weizmannia (Bacillus) Coagulans JBI-YZ6.3 on Gut Health and Fecal Microbiome Changes
Acronym: WIZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB-25-41
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Symptoms; Constipation; Gut Health; Gastrointestinal Function
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, placebo-controlled, crossover design. All participants will receive both interventions in a randomized order. Each participant will complete two 4-week supplementation periods, one with Weizmannia (Bacillus) coagulans JBI-YZ6.3 and one with placebo, separated by a 4-week washout period to minimize potential carryover effects.
  Participants will be randomly assigned to one of two treatment sequences: probiotic followed by placebo, or placebo followed by probiotic. Randomization will be stratified by sex, age, and body mass index. Both participants and study personnel will remain blinded to treatment assignment for the duration of the study.
  All participants will serve as their own control, allowing within-subject comparisons of gastrointestinal symptoms, stool characteristics, and fecal microbiome outcomes between the probiotic and placebo conditions.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weizmannia (Bacillus) coagulans JBI-YZ6.3 (Experimental)
  Interventions: Dietary Supplement: Weizmannia (Bacillus) coagulans JBI-YZ6.3
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Weizmannia (Bacillus) coagulans JBI-YZ6.3 — Participants will ingest Weizmannia (Bacillus) coagulans JBI-YZ6.3 daily for 4 weeks. The supplement will be provided in capsule form and consumed once daily with approximately eight ounces of water. Participants will be instructed to consume the supplement at the same time each day. If a dose is missed, participants will be instructed to take the missed dose the following day by splitting the dose into one capsule in the morning and one capsule in the evening. Supplementation will occur during one of two 4-week intervention periods as part of a randomized, double-blind, placebo-controlled crossover design.
  Arms: Weizmannia (Bacillus) coagulans JBI-YZ6.3
Dietary Supplement: Placebo — Participants will ingest a placebo consisting of microcrystalline cellulose in capsule form for 4 weeks. The placebo capsules will be identical in size, color, and appearance to the active supplement. Participants will consume the placebo once daily with approximately eight ounces of water at the same time each day. If a dose is missed, participants will be instructed to take the missed dose the following day by splitting the dose into one capsule in the morning and one capsule in the evening. Placebo supplementation will occur during one of two 4-week intervention periods as part of a randomized, double-blind, placebo-controlled crossover design
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of supplementation with Weizmannia (Bacillus) coagulans JBI-YZ6.3 on gastrointestinal health in healthy, physically active adults. The primary objective is to determine whether daily intake of this probiotic strain improves symptoms of constipation and related gastrointestinal function compared with placebo.

Approximately 30 healthy men and women aged 18 to 50 years will be enrolled in a randomized, double-blind, placebo-controlled, crossover trial. Participants will complete two 4-week supplementation periods, one with Weizmannia (Bacillus) coagulans JBI-YZ6.3 and one with placebo, separated by a 4-week washout period. The total duration of participation will be approximately 13 to 14 weeks, including screening and testing visits.

Gastrointestinal symptoms will be assessed at baseline and after each supplementation period using validated questionnaires, with particular focus on the constipation domain of the Gastrointestinal Symptom Rating Scale (GSRS). Secondary outcomes will include additional gastrointestinal symptom domains and markers of perceived gut comfort and function.

This study is designed to determine whether supplementation with Weizmannia (Bacillus) coagulans JBI-YZ6.3 produces clinically meaningful improvements in gastrointestinal symptoms in physically active adults compared with placebo.

DETAILED DESCRIPTION:
This study is designed to examine the effects of supplementation with Weizmannia (Bacillus) coagulans JBI-YZ6.3 on gastrointestinal health in healthy, physically active adults. Probiotic supplementation has been shown to influence gastrointestinal symptoms, intestinal barrier function, and microbial composition, but responses vary depending on strain, dose, and population. Weizmannia (Bacillus) coagulans JBI-YZ6.3 is a spore-forming probiotic strain that is highly stable and may survive gastric transit, allowing for potential effects on gut function and symptom perception. However, controlled clinical data in physically active adults are limited.

This study will employ a randomized, double-blind, placebo-controlled, crossover design to compare the effects of JBI-YZ6.3 with placebo. Approximately 30 healthy men and women aged 18 to 50 years will be recruited. All participants will be physically active and free of diagnosed gastrointestinal, metabolic, or inflammatory diseases.

After completing an online screening visit, eligible participants will complete two 4-week supplementation periods. During one period, participants will consume a daily dose of Weizmannia (Bacillus) coagulans JBI-YZ6.3, and during the other period they will consume a matched placebo. The order of treatments will be randomized. A 4-week washout period will separate the two supplementation phases to minimize any potential carryover effects. Participants will attend laboratory or virtual testing visits at the start and end of each supplementation period (weeks 0 and 4 of each phase).

Throughout the study, participants will be instructed to maintain their habitual diet, physical activity, and lifestyle behaviors, and to refrain from consuming additional probiotic or prebiotic supplements. Compliance with supplementation will be monitored by self-report and returned capsule counts.

The primary outcome of this study is the constipation domain of the Gastrointestinal Symptom Rating Scale (GSRS), a validated questionnaire used to assess gastrointestinal symptom severity. Secondary outcomes will include additional GSRS domains and other self-reported measures of gastrointestinal comfort and function.

Safety will be monitored throughout the study by collection of self-reported adverse events at each testing visit and via weekly check-ins during supplementation periods.

This study will determine whether daily supplementation with Weizmannia (Bacillus) coagulans JBI-YZ6.3 improves constipation-related symptoms and overall gastrointestinal health in physically active adults compared with placebo.

ELIGIBILITY:
Inclusion Criteria Ages of 18 - 50 years Average daily bloating score >5 on question 3 of the Modified daily Abdominal, Gas, and Bloating Questionnaire and/or bloating for >5 days during the past 14 days Body mass index (BMI) 18.5 - 29.9 kg/m2 (Inclusive) (Individuals >29.9 kg/m2, but <25% fat for men and <30% fat for women will be accepted into the study. The cohort average of body mass index will not exceed 29.9 kg/m2) Weight stable for the past three months (defined as less than a 5% variation in body mass over this time) Determined to be healthy through completion of a health history questionnaire Subject agrees to maintain their existing dietary patterns throughout the study period and to report to study investigators any changes particularly as they relate to probiotic-containing or fermented foods Subject agrees to refrain from alcohol, caffeine, and strenuous exercise for 24 hours prior to each test day.

Minimum baseline physical activity level (defined as at least 30 minutes of moderate intensity exercise at least 4 days per week for the past 3 months) Subject is willing and able to comply with the study protocol. Study participant is not currently enrolled in another clinical trial that involves the administration of some investigative agent Subject has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria Positive medical history and/or is currently being treated for some form of heart disease, cardiovascular disease Currently being treated for kidney disease, renal failure, or has dialysis performed on regular intervals Has liver disease or some form of clinically diagnosed hepatic impairment Diagnosed with having Type I or Type II diabetes (determined as fasting blood glucose > 126 mg/dL) Diagnosed with or is being treated for some form of thyroid disease Diagnosed with major affective disorder or other psychiatric disorder that required hospitalization in the prior year Diagnosed with some form of immune disorder (i.e., HIV/AIDS) History of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).

Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea) Participant has been treated for a gastrointestinal related disorder, complication, or disorder within the past 30 days Positive medical history for any neurological condition or neurological disease Diagnosed with or being treated for any endocrinological disorder or currently used any form of hormone replacement (prescribed/doctor ordered or not) Women with a history of hormone-related conditions such as endometriosis, fibroids, polycystic ovary syndrome Currently prescribed for the first time statin drugs (i.e., Lipitor, Livalo, Crestor, Zocor, etc.) within the past 6 months or has had their dosage or medication changed within the past 6 months Currently prescribed for the first time hypertension medication (i.e., Beta-blockers, ACE Inhibitors, Alpha blockers, Vasodilators, etc.) within the past 6 months or has had their dosage or medication changed within the past 6 months Current antibiotic use or other prescription or over-the-counter medications that may impact study outcomes Have a known sensitivity or allergy to any of the study products Blood donation in past 60 days Current smoker (average of > 1 pack per week within the past 3 months) or has quit within the past six months. This includes all forms of nicotine They plan major changes in lifestyle (i.e., diet, dieting, exercise level, travel, etc.) during the study Competitive athletes will be excluded History of alcohol or substance abuse in the 12 months prior to screening Current use of anabolic steroids (medically prescribed or otherwise) Receipt or use of an investigational product in another research study within 30 days of beginning the study protocol Report taking a probiotic or other dietary supplement know to impact digestion or gut function in the past 30 days Recent history (<3 months) of exercise training or weight loss (> 5%) Currently following a ketogenic or low carbohydrate diet within the past 30 days.

Women who are pregnant, planning to become pregnant, or lactating currently or within the past six months Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Constipation Score (Gastrointestinal Symptom Rating Scale) | Baseline and end of each 4-week supplementation period (Weeks 0 and 4 of each intervention period)
  Constipation will be assessed using the constipation domain of the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS is a validated 15-item questionnaire scored on a 7-point Likert scale, where higher scores indicate greater symptom severity. The constipation domain includes items related to hard stools, constipation, and sensation of incomplete bowel emptying. Scores will be compared between the Weizmannia (Bacillus) coagulans JBI-YZ6.3 and placebo conditions.

SECONDARY OUTCOMES:
Total GSRS Score | Baseline and end of each 4-week supplementation period
  Overall gastrointestinal symptom severity will be assessed using the total score of the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS includes 15 items rated on a 7-point Likert scale assessing gastrointestinal symptoms over the past week.
GSRS Symptom Domain Scores | Baseline and end of each 4-week supplementation period
  Individual GSRS domain scores for diarrhea, indigestion, abdominal pain, and reflux will be calculated and compared between the probiotic and placebo conditions.
Stool Consistency (Bristol Stool Chart) | Baseline, mid-intervention (Week 2 of each period), and end of each 4-week supplementation period
  Stool consistency will be assessed using the Bristol Stool Chart, which classifies stool form into seven categories ranging from hard pellets to watery stool. Scores will be compared between supplementation conditions.

OTHER OUTCOMES:
Resting Heart Rate | Baseline, mid-intervention (Week 2 of each period), and end of each 4-week supplementation period
  Resting heart rate will be measured using an automated blood pressure monitor after five minutes of seated rest.
Resting Blood Pressure | Baseline, mid-intervention (Week 2 of each period), and end of each 4-week supplementation period
  Resting blood pressure will be measured using an automated blood pressure monitor after five minutes of seated rest.

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data contain sensitive longitudinal biological and symptom information that cannot be reliably de-identified without compromising participant privacy.